CLINICAL TRIAL: NCT03414164
Title: In Vitro Effects of Procyanidine on Semen Parameters and DNA Fragmentation Index: a Prospective, Double-blind Trial
Brief Title: In Vitro Effects of Procyanidine on Semen Parameter and DFI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: Sohag University (Other)
Responsible Party: Principal Investigator, E.M. Kolibianakis, Associate Professor, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UHR-12
Record Dates: First submitted 2017-10-24; First posted 2018-01-29 (Actual); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Spermatogenesis and Semen Disorders; DNA Double Strand Break
MeSH Terms: interventions — procyanidin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- procyanidine group (Experimental)
  Interventions: Dietary Supplement: procyanidine
- control group (No Intervention)

INTERVENTIONS:
Dietary Supplement: procyanidine — natural antioxidants
  Arms: procyanidine group

SUMMARY:
Proanthocyanidins are a class of polyphenols found in a variety of plants that have antioxidant activity in vitro, which is stronger than vitamin C or vitamin E.

Several studies have been performed evaluating the administration of antioxidant therapy in the form of oral antioxidant supplementation or in vitro addition of antioxidant to culture media during assisted reproductive techniques (ART).

However, the impact of in vitro addition of proanthocyanidins to semen has not been studied yet. The research question evaluated in the current study was whether semen samples of infertile men supplemented or not with procyanidine immediately after their production, differ in semen parameters, sperm DFI.

ELIGIBILITY:
Inclusion Criteria:

* Infertility defined as:

  * At least twelve (12) months of non-achieving pregnancy despite unprotected sexual intercourse or six (6) months, if the female is > 35 years of age AND
  * At least two (2) semen analyses with at least one abnormal parameter (sperm concentration, motility and morphology), according to WHO 2010 criteria.
* Not on any type of infertility treatment for the last three (3) months
* Sperm concentration > 8 x 106/ml and semen volume at least 2.5 ml for technical reasons.
* Normal hormonal profile (TSH, FSH, LH, total testosterone, prolactin)
* Seminal white blood cells < 1 x 106/ml
* No abnormalities in scrotal ultrasound

Exclusion Criteria:

* Underlying genetic cause of infertility
* History of undescended testis (cryptorchidism)
* History of orchidectomy
* History of testicular cancer
* History of severe cardiac, hepatic or renal disease.
* History of endocrine disease (primary or secondary hypogonadism, hyperprolactinemia, thyroid disease, pituitary or adrenal disease)
* History of epididymo-orchitis, prostatitis, genital trauma, testicular torsion, inguinal or genital surgery
* History of systemic disease or treatment during the last three (3) months
* Positive sperm culture for Chlamydia or Ureaplasma urealyticum
* Female infertility factors
* Body mass index (BMI) > 30 kg/m2
* Participation in another interventional study and a likelihood of being unavailable for follow-up.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2017-04-29 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Progressive sperm motility | 3h after addition or not of procyanidine
  percentage (%) of decrease

SECONDARY OUTCOMES:
Sperm DNA fragmentation index | 3h after addition or not of procyanidine
  percentage (%) of decrease
Sperm morphology | 3h after addition or not of procyanidine
  percentage (%) of decrease
Sperm vitality | 3h after addition or not of procyanidine
  percentage (%) of decrease

CONTACTS AND LOCATIONS:
Locations (1):
- Stratis Kolibianakis, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided